CLINICAL TRIAL: NCT00528723
Title: Multicentre, Multinational, Randomised, Double Blind, Double Dummy, Active Drug Controlled, Parallel Group Study Design Clinical Trial of the Efficacy and Tolerability of Beclomethasone Dipropionate 250 mcg Plus Salbutamol 100 mcg in HFA pMDI Fixed Combination vs. Beclomethasone Dipropionate 250 mcg Plus Salbutamol 100 mcg in CFC pMDI (Clenil® Compositum 250) Fixed Combination in a 12-week Treatment Period of Adult Patients With Uncontrolled Asthma
Brief Title: Efficacy and Tolerability of Beclomethasone Plus Salbutamol in HFA pMDI Fixed Combination vs Beclomethasone Plus Salbutamol in CFC pMDI Fixed Combination in a 12-week Treatment Period of Adult Patients With Uncontrolled Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Nicolini Gabriele, Chiesi Farmaceutici
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MC/PR/033004/002/06; 2007-002816-25 (EudraCT Number)
Record Dates: First submitted 2007-09-11; First posted 2007-09-12 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Bronchial Asthma
Keywords: beclomethasone; as needed; salbutamol; wheezing
MeSH Terms: conditions — Asthma; Respiratory Sounds | interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): BDP/salbutamol HFA pMDI
  Interventions: Drug: salbutamol 100 mcg; Drug: BDP/salbutamol HFA pMDI
- B (Active Comparator): BDP/salbutamol CFC pMDI
  Interventions: Drug: salbutamol 100 mcg; Drug: BDP/salbutamol CFC pMDI

INTERVENTIONS:
Drug: salbutamol 100 mcg — To be used as needed for symptom relief
  Other Names: Ventolin®
Drug: BDP/salbutamol HFA pMDI — Patients assigned to BDP/salbutamol HFA pMDI will receive 2 puffs twice daily (morning and evening), for a total daily dose of BDP 1000 mcg/salbutamol 400 mcg, plus 2 puffs twice daily of alternative CFC placebo
  Arms: A
Drug: BDP/salbutamol CFC pMDI — Patients assigned to BDP/salbutamol CFC pMDI will receive 2 puffs twice daily (morning and evening), for a total daily dose of BDP 1000 mcg/salbutamol 400 mcg, plus 2 puffs twice daily of alternative HFA placebo
  Other Names: Clenil® Compositum 250
  Arms: B

SUMMARY:
The purpose of this trial is to verify if the test treatment BDP 250 mcg/salbutamol 100 mcg HFA pMDI fixed combination is non-inferior to BDP 250 mcg/salbutamol 100 mcg pMDI fixed combination given with the conventional CFC propellant (Clenil® Compositum 250, Chiesi Farmaceutici) in terms of Pulmonary Function (morning PEF).

DETAILED DESCRIPTION:
Asthma is a chronic inflammatory disorder of the airways and a serious public health worldwide problem, affecting people of all ages, with an estimate of 300 millions affected individuals.When uncontrolled, asthma can place severe limits on daily life, and can sometimes be fatal.

There are two major classes of inhaled therapy for the treatment of reversible obstructive airways disease: antinflammatory agents and bronchodilators. In particular, BDP 250 mcg plus salbutamol 100 mcg in fixed combination is an effective and safe method to control symptoms of persistent asthma in adults.

This study has been designed to compare the efficacy, safety and tolerability of a new BDP 250 mcg/salbutamol 100 mcg HFA pMDI fixed combination with the same CFC-formulated fixed combination, which is on the market from some decades.The HFA propelled product is developed to replace the CFC formulation already marketed according to the European Union's Committee for Proprietary Medicinal Products (CPMP) Note for Guidance (III/5378/93 - Final) in order to prevent from depletion of stratospheric ozone.

The primary objective of this trial is to demonstrate that the test treatment BDP 250 mcg/salbutamol 100 mcg HFA pMDI fixed combination is non-inferior to BDP 250 mcg/salbutamol 100 mcg pMDI fixed combination given with the conventional CFC propellant (Clenil® Compositum 250, Chiesi Farmaceutici) in terms of Pulmonary Function (morning PEF).

Given the aim of the study, the population to be monitored includes adult patients with persistent asthma according to the current guidelines. The treatment period will be preceded by a 2-week run-in period. Subjects satisfying all the inclusion and exclusion criteria will then enter the 12-week treatment period. Clinic visits will take place at the start and end of the run-in period, and after 2, 4, 8 and 12 weeks after randomisation.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained,
2. Male or female out-patients aged ³ 18 and < 65 years;
3. Uncontrolled asthma defined according to the GINA 2006 "Classification of Levels of Asthma Control". This definition includes the presence of two or more of the following features (in addition to the required range of FEV1): a) daytime asthma symptoms > twice a week; b) any limitation of activities; c) any nocturnal symptoms/awakening; b) need for reliever/rescue treatment > twice a week. These conditions are to be based on recent medical history and are to be confirmed in the 2-week run-in period;
4. Forced expiratory volume in the first second (FEV1) ³ 60% and < 80% of the predicted normal value;
5. Positive response to the reversibility test in the screening visit, defined as an increase of at least 12% (or, alternatively, of 200 mL) from pre-bronchodilator value in the measurement of FEV1 30 minutes following 4 puffs (4 ´ 100 µg) of inhaled salbutamol administered via pMDI. The reversibility test can be avoided in patients having a documented positive response in the previous 6 months;
6. Non-smokers or ex-smokers with a cumulative tobacco exposure less than 5 pack-years and who have stopped smoking since more than 1 year;
7. A co-operative attitude and ability to be trained to correctly use the pMDIs;
8. At the end of the 2-week run-in period, the condition of uncontrolled asthma (see inclusion criteria No. 3) is to be confirmed by reviewing the diary cards for run-in.

Exclusion Criteria:

1. Inability to carry out pulmonary function testing;
2. Diagnosis of Chronic Obstructive Pulmonary Disease (COPD;
3. History of near fatal asthma;
4. Evidence of severe asthma exacerbation or symptomatic infection of the airways in the previous 4 weeks;
5. Three or more courses of oral corticosteroids or hospitalisation due to asthma during the previous 6 months;
6. Patients who have been treated with an inhaled corticosteroid in the previous 4 weeks;
7. Patients who have been treated with nebulized, oral, intravenous or intramuscular corticosteroids in the past 8 weeks or depot injectable corticosteroids in the past 12 weeks;
8. Patients who have been treated with a long-acting β2-agonist (LABA) in the past 2 weeks;
9. Patients who have been treated with an oral β2-agonist in the past 48 hours;
10. Patients who have been treated with a short-acting β2-agonist (SABA) in the past 6 hours;
11. Patients who have been treated with nebulized bronchodilators in the past 2 weeks;
12. Patients who have been treated with anticholinergic medications (by any route) in the past 2 weeks;
13. Patients who have been treated with a xanthine derivative (by any route) in the past 4 weeks;
14. Patients who have been treated with an inhaled cromone or a leukotriene modifier in the past 4 weeks;
15. History or current evidence of heart failure, coronary artery disease, myocardial infarction, severe hypertension, cardiac arrhythmias;
16. Diabetes mellitus;
17. Percutaneous transluminal coronary angioplasty (PTCA) or coronary artery by-pass graft (CABG) during the previous six months;
18. Patients with an abnormal QTc interval value in the ECG test, defined as > 450 msec in males or > 470 msec in females;
19. Patients with a serum potassium value ≤ 3.5 mEq/L (or 3.5 mmol/L) and/or fasting serum glucose value ≥ 140 mg/dL (or 7.77 mmol/L);
20. Other haemodynamic relevant rhythm disturbances (including atrial flutter or atrial fibrillation with ventricular response, bradycardia (≤ 55 bpm), evidence of atrial-ventricular (AV) block on ECG of more than 1st degree;
21. Clinically significant or unstable concurrent diseases: uncontrolled hyperthyroidism, significant hepatic impairment, poorly controlled pulmonary (tuberculosis, active mycotic infection of the lung), gastrointestinal (e.g. active peptic ulcer), neurological or haematological autoimmune diseases;
22. Cancer or any chronic diseases with prognosis < 2 years;
23. Pregnant or lactating females or females at risk of pregnancy, i.e. those not demonstrating adequate contraception (i.e. barrier methods, intrauterine devices, hormonal treatment or sterilization).
24. History of alcohol or drug abuse;
25. Patients treated with monoamine oxidase inhibitors, tricyclic antidepressants or beta-blockers as regular use;
26. Allergy, sensitivity or intolerance to study drugs and/or study drug formulation ingredients;
27. Patients unlikely to comply with the protocol or unable to understand the nature, scope and possible consequences of the study;
28. Patients who received any investigational new drug within the last 12 weeks;
29. Patients who have been previously enrolled in this study;
30. At the end of the run-in period, patients will not be admitted to the treatment period in the case of an increase of FEV1 measured at the clinics at the end of the run-in period ³ 15% in respect of the pre-bronchodilator value measured at the start of the run-in period;
31. Patients with asthma exacerbations during the run-in period will also be excluded from the study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2007-11; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Mean value of morning PEF (daily measured by the patient) | last 2 weeks treatment

SECONDARY OUTCOMES:
Morning PEF daily measured by the patient at any other time point | last 2 weeks treatment
Evening PEF, and morning and evening FEV1 daily measured by the patient | all treatment period (12 weeks), at each two weeks
Pulmonary function parameters (FEV1, FVC, PEF and FEF25-75%) | clinic visits
Changes from pre-dosing of pulmonary function parameters measured at in the interval 0-60 minutes (pre-dose and 5, 15, 30 and 60 minutes post-dose); | baseline (visit 2) and end of treatment (visit 6)
Rates of asthma exacerbations (in total and by severity) | all treatment period, at each two weeks
Time to first asthma exacerbation | all treatment period, at each two weeks
Night-time and daytime use of relief salbutamol, and number of days (both day and night) without intake of salbutamol | all treatment period, at each two weeks
Nighttime and daytime symptoms scores, and number of symptoms-free days (both day and night) | all treatment period, at each two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Cremonesi, M D, Study Director — Chiesi Farmaceutici S.p.A.; Gabriele Nicolini, CPM, Study Director — Chiesi Farmaceutici S.p.A.; Luis Puente, Dr, Principal Investigator — Hospital General Universitario Gregorio Maranon, Madrid; Giorgio Walter Canonica, Prof., Principal Investigator — Ospedale S.Martino e Cliniche Universitarie Convenzionate, Genova, Italy; Igor Bereznyakov, Prof., Principal Investigator — Department of therapy of Kharkov Academy of Postgraduate Education, Kharkov, Ukraine
Locations (25):
- Italy (5):
  - Servizio di Fisiopatologia Respiratoria Diagnostica Allergologica e Biologia Respiratoria Endoscopica e Toracica U.O.C. di Pneumologia Ospedale Orlandi, Bussolengo, (vr)
  - Unità Dipartimentale di Fisiopatologia Respiratoria -Dipartimento di Medicina Interna e Specialità Mediche (DI.MI.) - Ospedale S. Martino e Cliniche Universitarie Convenzionate, Genova
  - Unità Operativa Complessa di Clinica fisiologica e Pneumologia - Dipartimento di Medicina Interna e Specialità Mediche (DI.MI.) - Ospedale S. Martino e Cliniche Universitarie Convenzionate, Genova
  - Dipartimento di Medicina Ambientale e Sanità Pubblica-Sede di Medicina del Lavoro Servizio di Fisiopatologia Respiratoria, Padua
  - Malattie dell'Apparato Respiratorio - Università degli Studi di Pisa Ospedale Cisanello, Pisa
- Russia (5):
  - City Clinical Hospital № 61, Pulmonology Department, Moscow
  - Central Clinical Hospital №1 OAO"RZD",Pulmonology Department, Moscow
  - Clinical Hospital № 2, Pulmonology Department, Yaroslavl
  - Clinical Hospital № 8, Pulmonology Department, Yaroslavl
  - Regional Clinical Hospital, Department of Therapeutics of Post Graduate, Yaroslavl Medical Academy, Yaroslavl
- Hospital General Universitario Gregorio Marañón, Madrid, Spain
- Ukraine (14):
  - Department of Therapy of Kharkov Medical Academy of Postgraduate Education City Multifield Clinical Hospital n° 25, Kharkiv
  - Pulmonological and Allergological Department of the Kharkov Regional Clinical Hospital, Kharkiv
  - Central Military Hospital of North Region. Pulmonological Department, Kharkiv
  - Department of propaedeutics of internal diseases #1. Kharkov State Medical University., Kharkiv
  - Pulmonological Department # 2 City Clinical Hospital # 13, Kharkiv
  - Pulmonological Department of the Institute of Therapy Ukrainian Academy of Medical Science, Kharkiv
  - Department of General Practice - Family Medecine Medical Academy of post-graduate education. City Clinical Hospital N° 17, Kharkiv
  - Department of Diagnostic, Therapy and Clinical Pharmacology of Lung Disease of the Institute of Phtisiology and Pulmonology Academy of Medical Sciences of the Ukraine, Kiev
  - Institute of Phthisiology and Pulmonology Acedemy of Medical Science of the Ukraine, Kiev
  - Pulmonology Department of the Institute of Phthisiology and Pulmonology AMS of the Ukraine, Kiev
  - Department of Pediatrics and laboratory diagnostics, Dniepropetrovsk State Medical Academy City Clinical Hospital No. 8. Pulmonology Department. 55, Krivoi Rog
  - General Therapy Clinic Central Military Clinical Hospital of Ministry of Defenses of Ukraine, Kyiv
  - Department of Hospital Therapy of Lugansk State Medical Institute, Luhansk
  - Department of Hospital Therapy, Lviv State Medical University named by Danylo Galytsky, Lviv Regional Clinical Hospital, Lviv

REFERENCES:
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=2007-002816-25